CLINICAL TRIAL: NCT01706926
Title: A Phase 2b Study to Evaluate the Efficacy and Safety of Mavrilimumab in Subjects With Moderate-to-Severe Rheumatoid Arthritis
Brief Title: A Study of Mavrilimumab in Subjects With Moderate-to-Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: MedImmune Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CD-IA-CAM-3001-1071
Record Dates: First submitted 2012-10-03; First posted 2012-10-15 (Estimated); Results first posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Mavrilimumab; CAM-3001
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — mavrilimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo matched to mavrilimumab (CAM-3001) injection subcutaneously every 2 weeks for 24 weeks in combination with stable dose of methotrexate (7.5 to 25 milligram [mg] per week) through oral or parenteral route.
  Interventions: Other: Placebo
- Mavrilimumab 30 mg (Experimental): Mavrilimumab (CAM-3001) 30 mg injection subcutaneously every 2 weeks for 24 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) through oral or parenteral route.
  Interventions: Biological: Mavrilimumab 30 mg
- Mavrilimumab 100 mg (Experimental): Mavrilimumab (CAM-3001) 100 mg injection subcutaneously every 2 weeks for 24 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) through oral or parenteral route.
  Interventions: Biological: Mavrilimumab 100 mg
- Mavrilimumab 150 mg (Experimental): Mavrilimumab (CAM-3001) 150 mg injection subcutaneously every 2 weeks for 24 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) through oral or parenteral route.
  Interventions: Biological: Mavrilimumab 150 mg

INTERVENTIONS:
Biological: Mavrilimumab 30 mg — Mavrilimumab (CAM-3001) 30 mg injection subcutaneously every 2 weeks for 24 weeks
  Other Names: CAM-3001
  Arms: Mavrilimumab 30 mg
Biological: Mavrilimumab 100 mg — Mavrilimumab (CAM-3001) 100 mg injection subcutaneously every 2 weeks for 24 weeks.
  Other Names: CAM-3001
  Arms: Mavrilimumab 100 mg
Biological: Mavrilimumab 150 mg — Mavrilimumab (CAM-3001) 150 mg injection subcutaneously every 2 weeks for 24 weeks.
  Other Names: CAM-3001
  Arms: Mavrilimumab 150 mg
Other: Placebo — Placebo matched to mavrilimumab (CAM-3001) injection subcutaneously every 2 weeks for 24 weeks.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of 3 subcutaneous doses of mavrilimumab compared with placebo in combination with methotrexate (MTX) in subjects with moderate-to-severe adult onset Rheumatoid Arthritis (RA).

DETAILED DESCRIPTION:
Despite the therapeutic improvements with recent biologic agents approved for rheumatoid arthritis, there is still significant unmet medical need for the treatment of subjects with this chronic disease to achieve a faster, more complete response, and higher rates of remission. The aim of the study is to explore the optimum dose of mavrilimumab for further clinical development and more fully investigate the efficacy and safety profile of mavrilimumab after longer drug exposure (that is, 24 weeks). The results of this study will form the basis for future clinical studies with mavrilimumab.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of adult onset Rheumatoid Arthritis (RA) in line with the protocol
* Moderately active disease in line with the protocol
* A pre-defined number of swollen joints in line with the protocol
* Inadequate response to one or more conventional disease-modifying anti-rheumatic drugs (DMARDs)
* No evidence of respiratory disease.

Exclusion Criteria:

* A rheumatic autoimmune disease other than RA, or significant systemic extra-articular involvement secondary to RA
* A history of, or current, inflammatory joint disease other than RA
* Previous treatment with the investigational drug
* Discontinuation of a biologic DMARD due to lack of efficacy
* Non-compliant concurrent medications
* Non-compliance with medical history criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marius Albulescu, MD, Study Director — MedImmune Ltd
Locations (42):
- Argentina (3):
  - Research Site, Ciudad Autonoma de Buenos Aire
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Chile (2):
  - Research Site, Santiago
  - Research Site, Viña del Mar
- Colombia (2):
  - Research Site, Barranquilla
  - Research Site, Bogotá
- Czechia (5):
  - Research Site, Bruntál
  - Research Site, Jihlava
  - Research Site, Ostrava - Trebovice
  - Research Site, Prague
  - Research Site, Zlín
- Research Site, Tallinn, Estonia
- Germany (3):
  - Research Site, Cologne
  - Research Site, Hildesheim
  - Research Site, Magdeburg
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Debrecen
- Poland (6):
  - Research Site, Gdynia
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (6):
  - Research Site, Barnaul
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Niška Banja
- Research Site, Durban, South Africa
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Santiago de Compostela
- Ukraine (5):
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Lutsk
  - Research Site, Vinnytsia

REFERENCES:
- [Derived] Burmester GR, McInnes IB, Kremer J, Miranda P, Korkosz M, Vencovsky J, Rubbert-Roth A, Mysler E, Sleeman MA, Godwood A, Sinibaldi D, Guo X, White WI, Wang B, Wu CY, Ryan PC, Close D, Weinblatt ME; EARTH EXPLORER 1 study investigators. A randomised phase IIb study of mavrilimumab, a novel GM-CSF receptor alpha monoclonal antibody, in the treatment of rheumatoid arthritis. Ann Rheum Dis. 2017 Jun;76(6):1020-1030. doi: 10.1136/annrheumdis-2016-210624. Epub 2017 Feb 17. PMID 28213566

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 420 participants were screened out of which 326 participants were randomized and received investigational product in the study.
Period: Overall Study
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Started | 81 | 81 | 85 | 79
Completed | 75 | 77 | 79 | 74
Not Completed | 6 | 4 | 6 | 5
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 2
Not completed — Other | 4 | 4 | 4 | 3

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) population analysis set included all participants in the treatment group corresponding to their randomized treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg | Total
Number analyzed (Participants) | 81 | 81 | 85 | 79 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (10.6) | 51.2 (11.6) | 50.8 (11.9) | 52.6 (10.3) | 51.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 70 | 70 | 67 | 282
  Male | 6 | 11 | 15 | 12 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score of 28 Joints Using C-Reactive Protein (DAS28 [CRP]) Score at Day 85
Description: DAS28 (CRP) calculated swollen joint count (SJC) and tender joint count (TJC) using the 28 joints, general health (GH) using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst), and CRP (milligram per liter [mg/L]). Total score range: 0-9.4, higher score= more disease activity. DAS28 (CRP) less than (<) 3.2 = low disease activity, greater than or equal to (>=) 3.2 to 5.1 = moderate to high disease activity and <2.6= remission. A Day 85 responder was defined as a participant who experienced more than 1.2 decrease from baseline in DAS28 (CRP) score at Day 85.
Time Frame: Baseline and Day 85
Population: The modified intent-to-treat (mITT) population analysis set included all participants in the treatment group corresponding to their randomized treatment group. Here "n" signifies participants who were evaluable for this measure for the specified time point for each arm, respectively.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
units on a scale
  Baseline (n=81, 81, 85, 79) | 5.78 (0.090) | 5.73 (0.104) | 5.91 (0.096) | 5.67 (0.086)
  Change at Day 85 (n=77, 76, 79, 78) | -0.68 (0.136) | -1.37 (0.136) | -1.64 (0.132) | -1.90 (0.136)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Analysis reported for change from baseline in DAS28 (CRP) at Day 85. An estimate of the treatment difference and its 95 percent (%) confidence interval (CI) was computed by means of repeated measures model, adjusted for baseline and including terms for treatment group, visit and treatment by visit interaction. Differences <0 favored mavrilimumab; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -0.69, 95% CI 2-sided [-1.06 to -0.31], Standard Error of Mean 0.193
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Analysis reported for change from baseline in DAS28 (CRP) at Day 85. An estimate of the treatment difference and its 95% CI was computed by means of repeated measures model, adjusted for baseline and including terms for treatment group, visit and treatment by visit interaction. Differences <0 favored mavrilimumab; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -0.96, 95% CI 2-sided [-1.33 to -0.58], Standard Error of Mean 0.190
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -1.22, 95% CI 2-sided [-1.60 to -0.84], Standard Error of Mean 0.193

2. Primary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 20 (ACR20) Responses at Day 169
Description: ACR20 was defined as >=20 percent (%) improvement, in: SJC and TJC and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and CRP.
Time Frame: Day 169
Population: The mITT population analysis set included all participants in the treatment group corresponding to their randomized treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
percentage of participants | 24.7 | 50.6 | 61.2 | 73.4
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Percent difference = 25.9, 95% CI 2-sided [11.5 to 40.3] — 95% unconditional exact CI was calculated using a test of treatment difference in proportion of responders using logistic regression with treatment as a factor. Differences greater than zero favored mavrilimumab
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Percent difference = 36.5, 95% CI 2-sided [22.5 to 50.5] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Percent difference = 48.7, 95% CI 2-sided [35.2 to 62.3] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and Day 169 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to Day 169
Population: The safety population included all participants who received any dose of investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
percentage of participants
  TEAEs | 46.9 | 50.6 | 42.4 | 54.4
  TESAEs | 1.2 | 4.9 | 5.9 | 2.5

4. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Any medically significant change in laboratory evaluations were recorded as adverse events. Following parameters were analyzed for laboratory examination: hematology (haemoglobin, absolute neutrophil count, leukocyte count, platelet count), serum chemistry (alanine transaminase, aspartate transaminase, bilirubin, gamma-glutamyl transferase), other serum chemistry (low-density lipoprotein cholesterol, triglycerides), and urinalysis.
Time Frame: Baseline up to Day 169
Population: The safety population included all participants who received any dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
participants
  Anemia | 1 | 1 | 0 | 0
  Eosinophilia | 0 | 0 | 1 | 0
  Leukocytosis | 2 | 0 | 0 | 0
  Lymphopenia | 0 | 0 | 0 | 1
  Neutropenia | 1 | 0 | 0 | 3
  Alanine aminotransferase increased | 0 | 1 | 1 | 1
  Aspartate aminotransferase increased | 0 | 1 | 1 | 0
  Gamma-glutamyltransferase increased | 0 | 1 | 0 | 0
  Hypertransaminasaemia | 0 | 0 | 2 | 2
  Dislipidaemia | 0 | 0 | 1 | 0
  Hypercholesterolaemia | 1 | 0 | 1 | 0
  Hyperlipidaemia | 0 | 2 | 0 | 3
  Hyperkalaemia | 0 | 0 | 0 | 1

5. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Vital sign assessments included blood pressure, pulse rate, temperature, weight and respiration rate. Vital signs abnormalities reported as TEAEs were reported.
Time Frame: Baseline up to Day 169
Population: The safety population included all participants who received any dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
participants
  Hypertension | 2 | 4 | 4 | 3
  Weight increased | 1 | 1 | 1 | 0
  Pyrexia | 0 | 1 | 0 | 0
  Hot flush | 0 | 0 | 1 | 0

6. Secondary Outcome: Percentage of Pulmonary Function Test Values Below Threshold Values at Day 169
Description: Pulmonary function testing were performed by spirometry to assess forced expiratory volume in 1 second (FEV1), forced expiratory volume in 6 second (FEV6), and forced vital capacity (FVC). FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FEV6 was the maximal volume of air exhaled in the six second of a forced expiration from a position of full inspiration. FVC was the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. The percentage of predicted values of these pulmonary function tests were calculated based on decreases from baseline and categorized as less than or equal to (=<) 15 percent (%), more than (>) 15 to =<20%, and >20%.
Time Frame: Day 169
Population: The safety population included all participants who received any dose of investigational product. Here "n" signifies participants who were evaluable for this measure for the specified threshold value mentioned parameter for each arm, respectively.
Measure: Number; unit: percent of pulmonary test values
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
percent of pulmonary test values
  FEV1 =<15% (n=42,67,75,75) | 97.6 | 98.5 | 96.0 | 89.3
  FEV1 >15 to 20% (n=42,67,75,75) | 0.0 | 0.0 | 1.3 | 6.7
  FEV1 >20% (n=42,67,75,75) | 2.4 | 1.5 | 2.7 | 4.0
  FEV6 =<15% (n=41,66,71,68) | 97.6 | 97.0 | 94.4 | 89.7
  FEV6 >15 to 20% (n=41,66,71,68) | 0.0 | 1.5 | 1.4 | 1.5
  FEV6 >20% (n=41,66,71,68) | 2.4 | 1.5 | 4.2 | 8.8
  FVC =<15% (n=42,67,75,75) | 97.6 | 98.5 | 94.7 | 94.7
  FVC >15 to 20% (n=42,67,75,75) | 0.0 | 0.0 | 1.3 | 2.7
  FVC >20% (n=42,67,75,75) | 2.4 | 1.5 | 4.0 | 2.7

7. Secondary Outcome: Dyspnea Score at Day 169
Description: Borg dyspnea scale is a validated participant reported outcome assessing participant's perceived difficulty in breathing (dyspnea). The scale ranges from 0 (nothing at all) to 10 (maximal difficulty). Higher scores indicate greater difficulty in breathing.
Time Frame: Day 169
Population: The safety population included all participants who received any dose of investigational product. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 41 | 65 | 73 | 74
units on a scale | 0.38 (0.62) | 0.22 (0.54) | 0.32 (0.73) | 0.28 (0.64)

8. Secondary Outcome: Oxygen Saturation Level at Day 169
Description: Oxygen saturation measured by pulse oximetry which measures the concentration of oxygen in the blood.
Time Frame: Day 169
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 40 | 65 | 73 | 74
percent saturation | 97.4 (1.4) | 97.4 (1.1) | 97.4 (1.1) | 97.3 (1.2)

9. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 50 (ACR50) Responses at Day 169
Description: ACR50 was defined as >=50% improvement, in: SJC and TJC and >=50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Day 169
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
percentage of participants | 12.3 | 28.4 | 25.9 | 40.5
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p = 0.013, Regression, Logistic; Percent difference = 16.0, 95% CI 2-sided [3.9 to 28.2] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.030, Regression, Logistic; Percent difference = 13.5, 95% CI 2-sided [1.8 to 25.3] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Percent difference = 28.2, 95% CI 2-sided [15.2 to 41.1] — [estimate comment as in outcome 2, analysis 1]

10. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 70 (ACR70) Responses at Day 169
Description: ACR70 was defined as >=70% improvement, in: SJC and TJC and >=70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Day 169
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
percentage of participants | 3.7 | 12.3 | 10.6 | 13.9
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p = 0.079, Fisher Exact; Percent difference = 8.6, 95% CI 2-sided [0.4 to 16.9] — 95% unconditional exact CI was calculated using the model of logit (response). p-value estimated from fisher's exact test
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.133, Fisher Exact; Percent difference = 6.9, 95% CI 2-sided [-0.8 to 14.6] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p = 0.026, Fisher Exact; Percent difference = 10.2, 95% CI 2-sided [1.5 to 18.9] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Change From Baseline in Continuous American College of Rheumatology (ACRn) Score at Day 169
Description: ACR score - continuous (ACRn) was defined as the minimum of the percentage improvement in TJC, SJC and the median of the percentage improvements in the other five components of the ACR criteria (participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; disability index of the HAQ; and CRP). Total score range was -100 to 100, where negative numbers indicated worsening and positive numbers indicated improvement.
Time Frame: Baseline up to Day 169
Population: The mITT population analysis set included all participants in the treatment group corresponding to their randomized treatment group. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 38 | 63 | 72 | 74
units on a scale | 13.25 (4.630) | 29.04 (3.828) | 30.24 (3.623) | 40.72 (3.644)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p = 0.009, Repeated measures model; Adjusted Mean difference = 15.79, 95% CI 2-sided [3.96 to 27.61], Standard Error of Mean 6.007 — An estimate of the treatment difference and its 95% CI was computed by means of repeated measures model, adjusted for baseline and including a treatment by visit interaction term. Differences <0 favored mavrilimumab
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.004, Repeated measures model; Adjusted mean difference = 16.99, 95% CI 2-sided [5.42 to 28.56], Standard Error of Mean 5.879 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = 27.47, 95% CI 2-sided [15.87 to 39.07], Standard Error of Mean 5.892 — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) Response by European League Against Rheumatism (EULAR) Category at Day 169
Description: DAS28 (CRP) response by EULAR category were used to measure individual response as none, moderate, and good, depending on the extent of change from baseline and the level of disease activity reached. Good response: change from baseline >1.2 with baseline DAS28 (CRP) <3.2; moderate response: change from baseline >1.2 with baseline DAS28 (CRP) >=3.2 to less than or equal to (=<) 5.1 or change from baseline >=0.6 to =< 1.2 with baseline DAS28 (CRP) >=3.2 to =<5.1; no response: change from baseline <0.6 or change from baseline >=0.6 and =<1.2 with baseline DAS28 (CRP) >5.1.
Time Frame: Day 169
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
percentage of participants
  No response | 65.4 (0.090) | 30.9 (0.104) | 28.2 (0.096) | 19.0 (0.086)
  Moderate response | 25.9 (0.136) | 35.8 (0.136) | 40.0 (0.132) | 41.8 (0.136)
  Good response | 8.6 | 33.3 | 31.8 | 39.2
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p < 0.001, Proportional odds analysis; Odds Ratio (OR) = 4.70, 95% CI 2-sided [2.56 to 8.80] — Odds ratio, 95% CI and p-value were was calculated using proportional odds analysis of response model including treatment as a factor. Odds ratios greater than (>) one favored mavrilimumab
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p < 0.001, Proportional odds analysis; Odds Ratio (OR) = 4.81, 95% CI 2-sided [2.64 to 8.92] — Odds ratio, 95% CI and p-value were was calculated using proportional odds analysis of response model including treatment as a factor. Odds ratios >one favored mavrilimumab
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Proportional odds analysis; Odds Ratio (OR) = 7.11, 95% CI 2-sided [3.85 to 13.40] — [estimate comment as in outcome 12, analysis 2]

13. Secondary Outcome: Percentage of Participants With DAS28 (CRP) Remission and Low Disease Activity at Day 169
Description: DAS28 (CRP) calculated SJC and TJC using the 28 joints, GH using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst), and CRP (mg/L). Total score range: 0-9.4, higher score= more disease activity. Remission was defined as less than 2.6 DAS28 (CRP) score. Low disease activity was defined as less than 3.2 DAS28 (CRP) score.
Time Frame: Day 169
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
percentage of participants
  DAS28 (CRP) Remission | 4.9 | 21.0 | 17.6 | 19.0
  Low Disease Activity | 8.6 | 33.3 | 31.8 | 41.8
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; DAS28 (CRP) remission: p-value estimated from fisher's exact test when number of placebo or active responders was less than 5; Test type: Superiority or Other; p = 0.004, Fisher Exact; Percent difference = 16.0, 95% CI 2-sided [6.0 to 26.1] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.014, Fisher Exact; Percent difference = 12.7, 95% CI 2-sided [3.3 to 22.1] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.007, Fisher Exact; Percent difference = 14.0, 95% CI 2-sided [4.2 to 23.9] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 30 mg; The analysis reported DAS28 (CRP) low disease activity response; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Percent difference = 24.7, 95% CI 2-sided [12.7 to 36.6] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 100 mg; The analysis reported DAS28 (CRP) low disease activity response; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Percent difference = 23.1, 95% CI 2-sided [11.5 to 34.8] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 150 mg; The analysis reported DAS28 (CRP) low disease activity response; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Percent difference = 33.1, 95% CI 2-sided [20.7 to 45.6] — [estimate comment as in outcome 2, analysis 1]

14. Secondary Outcome: Mean Change From Baseline in Swollen and Tender Joint Count at Day 169
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form, no swelling = 0, swelling =1. Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form, no tenderness = 0, tenderness = 1.
Time Frame: Baseline and Day 169
Population: The mITT population analysis set included all participants in the treatment group corresponding to their randomized treatment group. Here "n" signifies participants who were evaluable for this measure for the specified time point for each arm, respectively.
Measure: Mean (Standard Error); unit: joint count
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
joint count
  SJC: Baseline (n=81,81,85,79) | 14.44 (0.765) | 17.80 (1.126) | 16.82 (0.930) | 15.72 (0.795)
  SJC: Change at Day 169 (n=40,65,73,74) | -4.97 (0.932) | -10.65 (0.809) | -11.18 (0.771) | -11.96 (0.787)
  TJC: Baseline (n=81,81,85,79) | 26.26 (1.250) | 27.48 (1.553) | 26.96 (1.544) | 26.70 (1.284)
  TJC: Change at Day 169 (n=40,65,73,74) | -7.90 (1.447) | -15.14 (1.265) | -16.35 (1.207) | -18.32 (1.234)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Analysis reported for change from baseline in swollen joint count at Day 169; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -5.68, 95% CI 2-sided [-8.12 to -3.24], Standard Error of Mean 1.237 — An estimate of the treatment difference and its 95% CI was computed by means of repeated measures model, adjusted for baseline and including terms for treatment group, visit and treatment by visit interaction. Differences <0 favored mavrilimumab
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Analysis reported for change from baseline in swollen joint count at Day 169; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -6.21, 95% CI 2-sided [-8.60 to -3.82], Standard Error of Mean 1.211 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Analysis reported for change from baseline in swollen joint count at Day 169; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -7.00, 95% CI 2-sided [-9.40 to -4.59], Standard Error of Mean 1.219 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Mavrilimumab 30 mg; Analysis reported for change from baseline in tender joint count at Day 169; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -7.24, 95% CI 2-sided [-11.02 to -3.45], Standard Error of Mean 1.922 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Mavrilimumab 100 mg; Analysis reported for change from baseline in tender joint count at Day 169; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -8.45, 95% CI 2-sided [-12.16 to -4.74], Standard Error of Mean 1.884 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Mavrilimumab 150 mg; Analysis reported for change from baseline in tender joint count at Day 169; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -10.42, 95% CI 2-sided [-14.17 to -6.67], Standard Error of Mean 1.901 — [estimate comment as in outcome 14, analysis 1]

15. Secondary Outcome: Mean Change From Baseline in Patient Assessment of Pain at Day 169
Description: Participants rated the severity of arthritis pain on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS), where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Baseline and Day 169
Population: as for outcome 14
Measure: Mean (Standard Error); unit: mm
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
mm
  Baseline (n=81, 81, 85, 79) | 62.16 (2.093) | 62.65 (2.110) | 63.58 (2.034) | 62.35 (2.217)
  Change at Day 169 (n=40, 65, 73, 74) | -15.20 (3.006) | -23.14 (2.563) | -23.31 (2.446) | -26.53 (2.483)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p = 0.045, Repeated measures model; Adjusted mean difference = -7.94, 95% CI 2-sided [-15.72 to -0.17], Standard Error of Mean 3.950 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.037, Repeated measures model; Adjusted mean difference = -8.11, 95% CI 2-sided [-15.73 to -0.48], Standard Error of Mean 3.876 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p = 0.004, Repeated measures model; Adjusted mean difference = -11.32, 95% CI 2-sided [-19.00 to -3.65], Standard Error of Mean 3.899 — [estimate comment as in outcome 14, analysis 1]

16. Secondary Outcome: Mean Change From Baseline in Patient Global Assessment (PGA) of Disease Activity at Day 169
Description: Participants responded to a question, "Considering all the ways your arthritis affects you, how are you feeling today?" by using a 0 - 100 millimeter (mm) VAS, where 0 = very well and 100 = very poorly.
Time Frame: Baseline and Day 169
Population: as for outcome 14
Measure: Mean (Standard Error); unit: mm
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
mm
  Baseline (n=81, 81, 85, 79) | 64.86 (1.892) | 63.79 (2.074) | 63.71 (1.957) | 62.39 (2.099)
  Change at Day 169 (n=40, 65, 73, 74) | -20.21 (3.148) | -21.06 (2.685) | -22.40 (2.560) | -25.69 (2.600)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p = 0.837, Repeated measures model; Adjusted mean difference = -0.85, 95% CI 2-sided [-8.99 to 7.29], Standard Error of Mean 4.137 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.589, Repeated measures model; Adjusted mean difference = -2.19, 95% CI 2-sided [-10.18 to 5.79], Standard Error of Mean 4.058 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p = 0.180, Repeated measures model; Adjusted mean difference = -5.48, 95% CI 2-sided [-13.52 to 2.55], Standard Error of Mean 4.083 — [estimate comment as in outcome 14, analysis 1]

17. Secondary Outcome: Mean Change From Baseline in Physician Global Assessment of Disease Activity (MDGA) at Day 169
Description: Physician Global Assessment of Arthritis was measured by asking the physician to assess the participant's current arthritis disease activity by placing a vertical line on a 0 to 10 centimeter (cm) VAS, where 0 cm = very good and 10 cm = very bad.
Time Frame: Baseline and Day 169
Population: as for outcome 14
Measure: Mean (Standard Error); unit: cm
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
cm
  Baseline (n=81, 81, 85, 79) | 6.60 (0.168) | 6.60 (0.162) | 6.81 (0.144) | 6.42 (0.166)
  Change at Day 169 (n=40, 65, 73, 74) | -2.39 (0.305) | -3.81 (0.254) | -3.85 (0.241) | -3.95 (0.243)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -1.41, 95% CI 2-sided [-2.20 to -0.63], Standard Error of Mean 0.397 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -1.46, 95% CI 2-sided [-2.23 to -0.69], Standard Error of Mean 0.389 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted mean difference = -1.56, 95% CI 2-sided [-2.33 to -0.79], Standard Error of Mean 0.391 — [estimate comment as in outcome 14, analysis 1]

18. Secondary Outcome: Mean Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Day 169
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item was scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range from 0 to 3; where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline and Day 169
Population: as for outcome 14
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
units on a scale
  Baseline (n=81, 80, 85, 79) | 1.63 (0.054) | 1.52 (0.070) | 1.58 (0.056) | 1.58 (0.059)
  Change at Day 169 (n=40, 65, 73, 74) | -0.29 (0.081) | -0.37 (0.072) | -0.46 (0.068) | -0.55 (0.069)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p = 0.479, Repeated measures model; Adjusted mean difference = -0.08, 95% CI 2-sided [-0.29 to 0.14], Standard Error of Mean 0.108 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.124, Repeated measures model; Adjusted mean difference = -0.16, 95% CI 2-sided [-0.37 to 0.04], Standard Error of Mean 0.106 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p = 0.017, Repeated measures model; Adjusted mean difference = -0.26, 95% CI 2-sided [-0.47 to -0.05], Standard Error of Mean 0.107 — [estimate comment as in outcome 14, analysis 1]

19. Secondary Outcome: Ratio of Change From Baseline in C-Reactive Protein (CRP) at Day 169
Description: CRP is a substance produced by the liver that increases in the presence of inflammation in the body. The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement in underlying disease.
Time Frame: Baseline, Day 169
Population: The mITT population analysis set included all participants in the treatment group corresponding to their randomized treatment group. Here "N" (Number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 38 | 63 | 72 | 74
ratio | 1.2971 (83.3) | 0.8784 (102.8) | 0.5197 (287.4) | 0.5856 (153.3)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p = 0.017, Repeated measures model; Adjusted geometric mean ratio = 0.64, 95% CI 2-sided [0.45 to 0.92] — An estimate of the treatment difference and its 95% CI was computed by means of repeated measures model including terms for baseline as a continuous covariate and treatment as a factor was used for the analysis. Ratio <1 favored mavrilimumab
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted geometric mean ratio = 0.46, 95% CI 2-sided [0.32 to 0.66] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted geometric mean ratio = 0.44, 95% CI 2-sided [0.31 to 0.63] — [estimate comment as in outcome 19, analysis 1]

20. Secondary Outcome: Ratio of Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Day 169
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. The farther the red blood cells have descended, the greater the inflammatory response.
Time Frame: Baseline, Day 169
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 40 | 64 | 73 | 74
ratio | 0.89 (57.0) | 0.67 (56.4) | 0.62 (55.3) | 0.58 (61.0)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p = 0.003, Repeated measures model; Adjusted geometric mean ratio = 0.72, 95% CI 2-sided [0.58 to 0.89] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted geometric mean ratio = 0.68, 95% CI 2-sided [0.55 to 0.84] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p < 0.001, Repeated measures model; Adjusted geometric mean ratio = 0.61, 95% CI 2-sided [0.49 to 0.75] — [estimate comment as in outcome 19, analysis 1]

21. Secondary Outcome: Percentage of Participants With Simplified Disease Activity Index (SDAI) Remission at Day 169
Description: The SDAI was the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, patient global assessment and physician global assessment assessed on 0 - 10 cm VAS; and C-reactive protein (CRP) (milligram per deciliter [mg/dL]). The SDAI total score ranges from 0 to 86, where higher scores indicates greater affection due to disease activity. SDAI remission was defined as a score less than or equal to 3.3.
Time Frame: Day 169
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
percentage of participants | 1.2 (0.054) | 6.2 (0.070) | 2.4 (0.056) | 5.1 (0.059)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p = 0.210, Fisher Exact; Percent difference = 4.9, 95% CI 2-sided [-0.8 to 10.7] — 95% unconditional exact CI was calculated using the model of logit (response) with treatment as a factor. Differences >0 favored mavrilimumab
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 1.000, Fisher Exact; Percent difference = 1.1, 95% CI 2-sided [-2.9 to 5.1] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p = 0.207, Fisher Exact; Percent difference = 3.8, 95% CI 2-sided [-1.6 to 9.2] — [estimate comment as in outcome 21, analysis 1]

22. Secondary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) Remission at Day 169
Description: The CDAI was the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, patient global assessment and physician global assessment assessed on 0 - 10 cm VAS. The CDAI total score ranges from 0 to 76 where higher scores indicates greater affection due to disease activity. CDAI remission was defined as a score less than or equal to 2.8.
Time Frame: Day 169
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
percentage of participants | 1.2 (0.054) | 6.2 (0.070) | 3.5 (0.056) | 7.6 (0.059)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p = 0.210, Fisher Exact; Percent difference = 4.9, 95% CI 2-sided [-0.8 to 10.7] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.621, Fisher Exact; Percent difference = 2.3, 95% CI 2-sided [-2.3 to 6.9] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p = 0.062, Fisher Exact; Percent difference = 6.4, 95% CI 2-sided [0.0 to 12.7] — [estimate comment as in outcome 21, analysis 1]

23. Secondary Outcome: Percentage of Participants With American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Remission at Day 169
Description: ACR/EULAR remission was defined as swollen joint count (0-66), tender joint count (0-68), CRP (mg/dL) and participant global assessment (0-10) all less than or equal to one.
Time Frame: Day 169
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
percentage of participants | 0.0 (0.054) | 3.7 (0.070) | 1.2 (0.056) | 1.3 (0.059)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p = 0.245, Fisher Exact; Percent difference = 3.7, 95% CI 2-sided [-0.4 to 7.8] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 1.000, Fisher Exact; Percent difference = 1.2, 95% CI 2-sided [-1.1 to 3.5] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p = 0.494, Fisher Exact; Percent difference = 1.3, 95% CI 2-sided [-1.2 to 3.7] — [estimate comment as in outcome 21, analysis 1]

24. Secondary Outcome: Mean Change From Baseline in Functional Assessment of Chronic Illness Therapy-fatigue (FACIT-fatigue) at Day 169
Description: FACIT-F is a 13-item questionnaire questionnaire to measure the degree of fatigue experiences by participants in the previous 7 days. Participants scored each item on a 5-point scale: 0 (not at all) to 4 (very much). Larger the participant's response to the questions (with the exception of 2 negatively stated), greater was the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score) where higher sore represent less fatigue.
Time Frame: Baseline and Day 169
Population: as for outcome 14
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
units on a scale
  Baseline (n=79, 80, 84, 79) | 26.75 (0.824) | 28.91 (1.078) | 28.45 (0.998) | 27.82 (0.950)
  Change at Day 169 (n=40, 65, 73, 74) | 4.53 (1.225) | 5.72 (1.039) | 6.80 (0.988) | 8.45 (0.997)
Statistical Analysis 1: Comparison: Placebo vs Mavrilimumab 30 mg; Test type: Superiority or Other; p = 0.463, Repeated measures model; Adjusted mean difference = 1.18, 95% CI 2-sided [-1.99 to 4.35], Standard Error of Mean 1.608 — An estimate of the treatment difference and its 95% CI was computed by means of repeated measures model, adjusted for baseline and including terms for treatment group, visit and treatment by visit interaction. Differences >0 favored mavrilimumab
Statistical Analysis 2: Comparison: Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.151, Repeated measures model; Adjusted mean difference = 2.27, 95% CI 2-sided [-0.83 to 5.37], Standard Error of Mean 1.574 — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Mavrilimumab 150 mg; Test type: Superiority or Other; p = 0.014, Repeated measures model; Adjusted mean difference = 3.92, 95% CI 2-sided [0.81 to 7.02], Standard Error of Mean 1.578 — [estimate comment as in outcome 24, analysis 1]

25. Secondary Outcome: Serum Concentrations of Mavrilimumab
Description: Serum concentrations after multiple subcutaneous doses of mavrilimumab were calculated for each cohort (30mg, 100mg and 150mg). Geometric coefficient of variation at Baseline for cohorts 30mg and 150mg were calculated as the negligible mean value was observed.
Time Frame: Baseline, Day 8, 15, 29, 85, 141, and 169
Population: The pharmacokinetic (PK) population included all participants who received mavrilimumab and for whom serum concentrations of mavrilimumab were available for PK data analyses. Here "n" signifies participants who were evaluable for the specified time point for each arm, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 85 | 79
nanogram per milliliter
  Baseline (n=80, 85, 79) | 0.00 (894.4) | 0.00 (NA) — Geometric coefficient of variation could not be calculated as mean and geometric mean were zero at this time point. | 0.00 (862.0)
  Day 8 (n=78, 83, 78) | 617.49 (111.8) | 3563.31 (49.3) | 6087.06 (43.4)
  Day 15 (n=78, 84, 78) | 154.60 (194.2) | 2479.96 (52.1) | 4616.35 (42.6)
  Day 29 (n=77, 85, 76) | 217.67 (248.3) | 4503.97 (54.8) | 7843.66 (42.9)
  Day 85 (n=74, 81, 77) | 201.57 (162.8) | 6538.22 (52.7) | 13213.93 (50.1)
  Day 141 (n=67, 75, 71) | 258.77 (136.9) | 2932.80 (75.6) | 9241.31 (52.1)
  Day 169 (n=63, 73, 74) | 348.97 (141.2) | 5282.37 (62.0) | 9178.47 (56.6)

26. Secondary Outcome: Percentage of Participants Exhibiting Anti-Drug Antibodies (ADAs) to Mavrilimumab at Any Visit
Description: Immunogenicity assessment included determination of anti-drug (mavrilimumab) antibodies in serum samples. ADA detection measured by using electrochemiluminescence assays.
Time Frame: Day 1 to Day 169
Population: The immunogenicity population included all participants who received at least 1 dose of mavrilimumab and for whom at least one serum sample for immunogenicity testing was available.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Number analyzed (Participants) | 81 | 81 | 85 | 79
percentage of participants | 2.5 | 16.0 | 3.5 | 0.0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 169
Arm/Group | Placebo | Mavrilimumab 30 mg | Mavrilimumab 100 mg | Mavrilimumab 150 mg
Serious Adverse Events (participants affected / at risk) | 1/81 | 4/81 | 5/85 | 2/79
Other Adverse Events (participants affected / at risk) | 38/81 | 41/81 | 36/85 | 43/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | Mavrilimumab 30 mg (N=81) | Mavrilimumab 100 mg (N=85) | Mavrilimumab 150 mg (N=79)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | Mavrilimumab 30 mg (N=81) | Mavrilimumab 100 mg (N=85) | Mavrilimumab 150 mg (N=79)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 6 (6) | 3 (3) | 1 (1) | 4 (4)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 4 (5) | 3 (4) | 6 (6)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chemical poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (3) | 2 (2) | 0 (0)
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 5 (5) | 4 (4) | 6 (8)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dyssomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 4 (4) | 4 (5) | 3 (3)
Venous insufficiency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Non-compartmental analyses was not performed for pharmacokinetics parameters due to limited sampling schedule

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.